CLINICAL TRIAL: NCT04576546
Title: Use of Inositols Within IVF Protocols to Reduce Gonadotropin Administration
Brief Title: Inositols and FSH in IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MI_DCI_FSH
Record Dates: First submitted 2020-09-30; First posted 2020-10-06 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Amount of FSH Units During Ovarian Stimulation Protocols
MeSH Terms: interventions — Inositol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- comparator group (Active Comparator): myo-inositol treatment
  Interventions: Dietary Supplement: Myo-inositol
- study group (Experimental): D-chiro-inositol treatment
  Interventions: Dietary Supplement: D-chiro-inositol

INTERVENTIONS:
Dietary Supplement: D-chiro-inositol — Supplementation of D-chiro-inositol (1000 mg/die), starting at least 4 weeks before rFSH administration
  Arms: study group
Dietary Supplement: Myo-inositol — Supplementation of myo-inositol (4 g/die), starting at least 4 weeks before rFSH administration
  Arms: comparator group

SUMMARY:
Ovarian hyperstimulation syndrome (OHSS), although quite uncommon, represents the most serious complication of ovulation induction during in-vitro fertilization (IVF) protocols. The syndrome is triggered by exaggerated ovarian response to gonadotropins, which eventually leads to pathological manifestations that range from mild symptoms, such as abdominal discomfort, to life-threatening complications in the most severe cases. Prevention is paramount during fertilization programs and requires assessment of risk factors and close monitoring of risk markers. Clinicians quite generally consider unusually elevated estrogen levels as both indicator for OHSS and one possible etiological factor. In this scenario, myo-inositol (MYO) treatment proved to reduce the amount of FSH units and the duration of the stimulation protocol, decreasing the risk of OHSS onset. On the other hand, inconclusive evidence is available about the effect of D-chiro-inositol (DCI) supplementation within assisted reproductive treatments. The aim of the proposed pilot study is to assess the effect of DCI supplementation on the doses of FSH used in IVF-ET protocols, also with respect to MYO treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing IVF-ET procedure
* HOMA-IR index < 2.0
* AMH in the range 1.0 - 2.0 ng/ml

Exclusion Criteria:

* History of cancelled IVF cycles
* BMI < 20 kg/m2 or ≥ 30 kg/m2
* Diagnosis of PCOS
* Thyroid diseases
* Presence of co-morbidities

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 300 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
FSH units/retrieved oocyte | 1 day (single time-point at ovulation)
  number of IU of recombinant FSH administered, normalized on the number of oocytes retrieved during the pick-up

SECONDARY OUTCOMES:
Total FSH (IU) | 1 day (single time-point at ovulation)
  total number of FSH IU used in the stimulation protocol
Duration of the stimulation | 1 day (single time-point at ovulation)
  Number of days of the stimulation protocol till pick-up
number of viable oocytes | 1 day (single time-point at oocyte pick-up)
  number of retrieved oocytes eligible for fortilization
oocyte quality | 1 day (single time-point at oocyte pick-up)
  classification of oocyte quality before fertilization
embryo quality | 1 day (single time-point at embryo transfer)
  evaluation of the quality of embryos after fertilization, before transfer

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Alma Res, Roma, Italy

IPD SHARING:
Plan to Share IPD: No